CLINICAL TRIAL: NCT00690859
Title: Evaluation of Predictor Factors of Recurrence in Bipolar Disorder in Spain
Brief Title: Predictors of Recurrence in Bipolar Disorder in Spain
Acronym: PREBIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Teresa Díez, PhD, Local MC Neuroscience Therapeutic Area Manager, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NES-DUM-2007/1
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2009-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorders; Predictors of recurrence
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Ambulatory bipolar I and II patients, clinically stabilized for at least the two months prior to recruitment and who had at least one acute episode (depressive, manic, hypomanic or mixed) within the year prior to recruitment.

SUMMARY:
Observational, prospective (1 year follow up), multicenter, non-interventional open label study in order to assess the factors that predict onset of mood disorders episodes (depression, mania, hypomania and mixed) in stabilized patients with bipolar disorder I or II in Spain. Other objectives are

1. to describe the clinical course of illness in a cohort of patients with TB I or II: duration, severity, polarity and seasonality
2. to describe clinical and functional situation of patients during the different phases, evaluating prognostic meaning of subsyndromal symptoms
3. to evaluate the economical impact on health service of these patients (hospitalization, primary care, treatments…).

Target population is ambulatory bipolar I and II patients, clinically stabilized for at least the two months prior to recruitment and who had at least one acute episode (depressive, manic, hypomanic or mixed) within the year prior to recruitment. The primary endpoint is the onset of mood disorders episodes (depression, mania, hypomania and mixed) during the follow-up period and evaluation of which factors predict onset of mood episodes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of Bipolar Disorder I or II (DSM-IV-TR)
* Patients Stabilized from at least 2 months who had a mood disorder episode (depression, mania, hypomania or mixed) in the last year.
* To be attended by a psychiatric specialist

Exclusion Criteria:

* Inability to participate in the study
* To have taken part in other study in the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory bipolar I and II patients, clinically stabilized for at least the two months prior to recruitment and who had at least one acute episode (depressive, manic, hypomanic or mixed) within the year prior to recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 595 (Actual)
Dates: Start 2007-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Onset of mood disorders episodes (depression, mania, hypomania and mixed) during the 1 year follow-up period | Every three months
Evaluation of the factors that predict onset of mood episodes (depression, mania, hypomania and mixed) | Every three months

SECONDARY OUTCOMES:
Evaluation of factors that can predict functional outcomes | Every three months
Description of Health services utilization (hospitalisations, primary care, treatments..) | Every three months

CONTACTS AND LOCATIONS:
Locations (49):
- Spain (49):
  - Research Site, Victoria, Alava
  - Research Site, Elda, Alicante
  - Research Site, Torrevieja, Alicante
  - Research Site, El Ejido, Almeria
  - Research Site, Langreo, Austurias
  - Research Site, Manresa, Barcelona
  - Research Site, Sabadell, Barcelona
  - Research Site, Terrassa, Barcelona
  - Research Site, Vilafranca del Penedès, Barcelona
  - Research Site, Coria, Caceres
  - Research Site, El Puerto de Santa María, Cadiz
  - Research Site, Santander, Cantabria
  - Research Site, Donostia / San Sebastian, Guipuzcoa
  - Research Site, Andújar, Jaen
  - Research Site, Conxo, La Coruna
  - Research Site, Calahorra, La Rioja
  - Research Site, Arucas, Las Palmas
  - Research Site, Banaderos, Las Palmas
  - Research Site, Arganda, Madrid
  - Research Site, Fuenlabrada, Madrid
  - Research Site, Torrejón de Ardoz, Madrid
  - Research Site, Velez, Malaga
  - Research Site, Vigo, Pontevedra
  - Research Site, Gijón, Principality of Asturias
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Mairena del Aljarafe, Sevilla
  - Research Site, Foios, Valencia
  - Research Site, Sagunto, Valencia
  - Research Site, Vilanova, Valencia
  - Research Site, Barakaldo, Vizacaya
  - Research Site, Zalla, Vizcaya
  - Research Site, Zamudio, Vizcaya
  - Research Site, Toro, Zamora
  - Research Site, Barcelona
  - Research Site, Burgos
  - Research Site, Granada
  - Research Site, Jaén
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Murcia
  - Research Site, Ourense
  - Research Site, Palma de Mallorca
  - Research Site, Salamanca
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
  - Research Site, Valencia
  - Research Site, Valladolid
  - Research Site, Zaragoza